CLINICAL TRIAL: NCT02743858
Title: A Prospective Surveillance Program for Assessment and Treatment of Breast Cancer-Related Lymphedema After Axillary Lymph Node Dissection
Brief Title: Lymphedema Surveillance Study
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 16-220
Record Dates: First submitted 2016-04-08; First posted 2016-04-19 (Estimated); Last update posted 2025-07-01 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Lymphedema
Keywords: Lymphedema; Surveillance Program; Axillary Lymph Node Dissection; 16-220
MeSH Terms: conditions — Breast Neoplasms; Lymphedema | interventions — Body Mass Index; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — breast tissue

GROUPS / COHORTS (3):
- Patients who consent for ALND: In patients treated with ALND, bilateral arm measurements will be obtained using the Perometer (Model 350 NT Perometer, Per-System) circumferential arm measurements with elastic tape taken at 4-cm intervals from the wrist to the shoulder & the L-Dex U400 (Impedimed, Brisbane, Australia) for bioimpedance measurements. Measurements will be performed at baseline (prior to surgery), post-operatively (after surgery) & at scheduled timepoints of 6 months, 12 months, 18 months, & 24 months after surgery for a total of 2 years. For a patient who is diagnosed with lymphedema at ≥ 13 months after surgery, surveillance will continue for an additional 12 months after [lymphedema] diagnosis, & total surveillance time may exceed 2 years. Height & weight will be obtained for each patient at baseline & at each scheduled visit for the purpose of calculating BMI. All patients will complete the ULL-27 (upper limb lymphedema) quality-of-life questionnaire at baseline & at each scheduled visit.
  Interventions: Other: Bilateral arm measurements; Other: Body mass index (BMI); Behavioral: Quality of Life Questionnaire
- Patients treated with SLNB alone: Study requirements which include arm measurements, height and weight and completion of a questionnaire at a single long-term follow-up timepoint, will be explained to the patient
  Interventions: Other: Bilateral arm measurements; Other: Body mass index (BMI); Behavioral: Quality of Life Questionnaire
- ALND Translational Study Patients: Patients will also be counseled about blood draws, which will include withdrawal of up to 20 mL of blood. Patients who are eligible and agree to participate will sign a consent form. Arm measurements, height and weight, blood draw (if applicable), and baseline questionnaire will be performed at first contact if possible, or at a follow-up scheduled visit prior to surgery.
  Interventions: Other: Bilateral arm measurements; Other: Body mass index (BMI); Behavioral: Quality of Life Questionnaire; Other: Blood draw

INTERVENTIONS:
Other: Bilateral arm measurements — Pts treated with ALND, bilateral arm measurements will be obtained using the Perometer (Model 350 NT Perometer, Per-System) circumferential arm measurements with elastic tape taken at 4-cm intervals from the wrist to the shoulder & the L-Dex U400 (Impedimed, Brisbane, Australia) for bioimpedance measurements. Measurements will be performed before surgery, post-operatively & at timepoints of 6,12,18, & 24 months after surgery for 2 years will be obtained using the Perometer (Model 350 NT Perometer, Per-System) for bioimpedance measurements. Pts who have not yet developed lymphedema by 2 years, an additional measurement at approx 3 years post-surgery will be performed. If pt is diag with lymphedema at the 3-year visit, she will be asked to continue on study for an additional year. Pts treated with SLNB alone, following re-consent, a long-term follow-up volumetric arm measurement will be obtained using the perometer & circumferential arm measurements at a minimum of 2 years post-surgery.
Other: Body mass index (BMI) — Height and weight will be obtained for each patient at baseline and at each scheduled visit for the purpose of calculating BMI. BMI will be correlated with the presence of inflammatory biomarkers in the tissue, as well as with lymphedema development.
Behavioral: Quality of Life Questionnaire
Other: Blood draw — Patients enrolled in the translational study (Cohort 3) will undergo blood draws for serum collection preoperatively and 12-24 months postoperatively to test for FGF2, IL4, IL10, TGFB, Leptin, IL6, and CRP. At both timepoints, up to 20 mL of blood will be collected.
  Groups: ALND Translational Study Patients

SUMMARY:
This study is being done to find out how many women develop lymphedema after an axillary lymph node dissection. The investigators also want to look for reasons why some women get lymphedema and others don't. Specifically, the investigators want to do tests on the breast tissue that is removed at the time of surgery to see if they can identify inflammation in the breast tissue, which may increase a woman's risk for lymphedema. The investigators will also ask the patient to answer questions to see how much their quality of life is affected by lymphedema, and whether this study can help women by detecting lymphedema earlier.

ELIGIBILITY:
Inclusion Criteria:

* Female breast cancer patients over the age of 18
* Patients consenting for unilateral axillary lymph node dissection (ALND) (prior history of sentinel lymph node biopsy allowed if <6 months from consent)
* Patients consenting for unilateral sentinel lymph node biopsy (SLNB) and possible ALND are eligible for initial entry into the study, but will become ineligible if ALND is not performed
* Initially consented patients, treated with SLNB alone, who were originally considered ineligible to continue on study, will be approached for re-enrollment
* Patients who self-identify as Black or White consenting for unilateral ALND or possible ALND will be approached for enrollment onto translational study (Cohort 3)

Exclusion Criteria:

* Male breast cancer patients
* Patients consenting for bilateral axillary surgery
* Patients with prior history of surgical excision of one or more axillary lymph nodes or SLNB, performed >6 months from date of consent
* Patients with prior history of ALND
* Patients with no breast surgery performed at MSK

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MSK clinics
Sampling Method: Non-Probability Sample
Enrollment: 1250 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
number of incidences of lymphedema | 2 year
  as defined by perometry using rigorous measurement protocols. Bilateral arm measurements will be obtained using the Perometer (Model 350 NT Perometer, Per-System) and the L-Dex U400 (Impedimed, Brisbane, Australia) for bioimpedance measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Barrio, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Consent only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent only), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Consent only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Consent only), Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/